CLINICAL TRIAL: NCT04420221
Title: A Phase I/II, Observer-blind, Randomised, Placebo-controlled Study to Assess Safety, Immunogenicity and Efficacy of GSK S. Aureus Candidate Vaccine When Administered to Healthy Adults (Dose-escalation) and to Adults 18 to 64 Years of Age With a Recent S. Aureus Skin and Soft Tissue Infection (SSTI)
Brief Title: Safety, Immunogenicity and Efficacy of GSK S. Aureus Candidate Vaccine (GSK3878858A) When Administered to Healthy Adults (Dose-escalation) and to Adults 18 to 64 Years of Age With a Recent S. Aureus Skin and Soft Tissue Infection (SSTI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 208833; 2021-006215-29 (EudraCT Number)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Infections, Soft Tissue
Keywords: S. aureus; skin and soft tissue infection; first time in human; S. aureus vaccine
MeSH Terms: conditions — Soft Tissue Infections; Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1 Dose-escalation Safety Lead-in Epoch: Half dose Non-Adjuvant (Non-Adj) (Experimental): Participants received 1 dose of the half dose formulation of the vaccine on Day 1.
  Interventions: Biological: Sa-5Ag half dose non-adjuvanted
- Group 2 Dose-escalation Safety Lead-in Epoch: Full dose Non-Adj (Experimental): Participants received 1 dose of the full dose formulation of the vaccine on Day 1.
  Interventions: Biological: Sa-5Ag full dose non-adjuvanted
- Group 3 Dose-escalation Safety Lead-in Epoch: Half dose Adj (Experimental): Participants received 1 dose of the half dose formulation of the vaccine with adjuvant on Day 1.
  Interventions: Biological: Sa-5Ag half dose adjuvanted
- Group 4 Dose-escalation Safety Lead-in Epoch: Full dose Adj (Experimental): Participants received 2 doses of the full dose formulation of the vaccine with adjuvant on Day 1 and Day 61.
  Interventions: Biological: Sa-5Ag full dose adjuvanted
- Dose-escalation Safety Lead-in Epoch: Placebo (Placebo Comparator): Participants received matching placebo on Day 1 for Group 1, Group 2 and Group 3, and on Day 1 and Day 61 for Group 4 of the escalation epoch.
  Interventions: Biological: Placebo
- Proof of Principle (PoP): Full dose Adj (Experimental): Participants were randomized to receive 2 doses of the full dose formulation of the vaccine with adjuvant on Day 1 and Day 61.
  Interventions: Biological: Sa-5Ag full dose adjuvanted
- PoP: Placebo (Placebo Comparator): Participants were randomized to receive 2 doses of placebo on Day 1 and Day 61.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Sa-5Ag half dose non-adjuvanted — 1 dose of Sa-5Ag (5 antigens of S. aureus) half dose, non-adjuvanted at Day 1, administered intramuscularly.
  Arms: Group 1 Dose-escalation Safety Lead-in Epoch: Half dose Non-Adjuvant (Non-Adj)
Biological: Sa-5Ag full dose non-adjuvanted — 1 dose of Sa-5Ag (5 antigens of S. aureus) full dose, non-adjuvanted at Day 1, administered intramuscularly.
  Arms: Group 2 Dose-escalation Safety Lead-in Epoch: Full dose Non-Adj
Biological: Sa-5Ag half dose adjuvanted — 1 dose of Sa-5Ag (5 antigens of S. aureus) half dose, adjuvanted at Day 1, administered intramuscularly.
  Arms: Group 3 Dose-escalation Safety Lead-in Epoch: Half dose Adj
Biological: Sa-5Ag full dose adjuvanted — A series of 2 doses of S. aureus candidate vaccine (Sa-5Ag full dose adjuvanted) given approximately 2 months apart (Days 1 and 61), administered intramuscularly.
  Arms: Group 4 Dose-escalation Safety Lead-in Epoch: Full dose Adj; Proof of Principle (PoP): Full dose Adj
Biological: Placebo — One dose of placebo (saline solution for injection/ vial or prefilled syringe) at Day 1 for placebo Groups 1 to 3 (Dose-escalation epoch) and a series of 2 doses of placebo given approximately 2 months apart (Days 1 and 61) for placebo Group 4 (Dose-escalation epoch) and Group PoP: Placebo, administered intramuscularly.
  Arms: Dose-escalation Safety Lead-in Epoch: Placebo; PoP: Placebo

SUMMARY:
The study evaluates the safety, immunogenicity, and efficacy of the GSK S. aureus candidate vaccine (GSK3878858A) when administered to two groups: healthy adults (dose-escalation phase) and adults aged 18 to 64 years with a recent S. aureus skin and soft tissue infection (SSTI). In the dose-escalation safety lead-in phase, the safety and immunogenicity of four different vaccine compositions are assessed in healthy adults. Once safety has been established in this phase, the second phase, known as the proof of principle (PoP) phase, will assess the safety, immunogenicity, and efficacy of the final vaccine composition in adults with a recent SSTI.

ELIGIBILITY:
Inclusion Criteria:

All participants must satisfy all the following criteria at study entry:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* Written or witnessed informed consent obtained from the participant prior to performance of any study specific procedure.
* Participant satisfying screening requirements.
* Participants who, after the nature of the study has been explained to them, have shown adequate comprehension of the study procedures and knowledge of study.
* A male or female
* Dose escalation and safety lead-in phase: Aged between 18 and 50 years of age, inclusive, at the time of first vaccination.
* PoP phase: Aged between 18 and 64 years of age, inclusive, at the time of first vaccination.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant:
* has practiced adequate contraception for 30 days prior to vaccination,
* has a negative pregnancy test on the day of enrolment, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Additional inclusion criteria only for participants to be enrolled in the dose-escalation safety lead-in screening epoch:

- Healthy participants as established by medical history, clinical examination and laboratory assessment.

Additional inclusion criteria only for participants to be enrolled in the PoP screening epoch:

- Healthy participants as established by medical history and clinical examination before entering into the study with an ongoing SSTI suspected to be caused by S. aureus, as diagnosed by investigator (before randomization participants have to be treated until clinical resolution of culture confirmed SSTI caused by S. aureus). SSTI must be amenable to microbiological culturing per standard clinical practice (i.e. recovery of drainage sample from abscess or suppurative cellulitis).

OR

- Healthy participants as established by medical history and clinical examination before entering into the study with an ongoing S. aureus SSTI (i.e. S. aureus is the most likely cause), as confirmed by a S. aureus positive culture performed outside the study procedures and not earlier than 30 days prior to Informed Consent Form signature. Before randomisation participants have to be treated until clinical resolution of the culture confirmed SSTI caused by S. aureus. These participants will be enrolled whether they have or have not already started specific treatment of the infection. In case they have not started the treatment, this will be then given in compliance with the standard medical practice for the management of S. aureus SSTIs and the choice and judgment of the most appropriate treatment will be applied by the investigator, outside the study procedures.

Exclusion Criteria:

All participants at study entry

* Body mass index (BMI) >40 kg/m2
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine
* Hypersensitivity to latex
* Recurrent history of uncontrolled neurological disorders or seizures
* History of potential immune-mediated disease (pIMD)
* Clinical conditions that in the investigator's opinion represent a contraindication to intramuscular vaccination and blood draws
* Known bleeding diathesis or any condition that may be associated with a prolonged bleeding time
* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study vaccine(s) within 30 days before the first dose of study vaccine(s)/placebo (Day -29 to Day 1), or during the study period
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine/placebo dose
* Cytotoxic therapy (e.g., medications used during cancer chemotherapy)
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab)
* Administration of immunoglobulins and/or any blood products or plasma derivatives within 3 months before the first dose of study vaccine or during the study period
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 15 days before the first dose and ending 15 days after the last dose of vaccine(s) administration with the exception of any non-adjuvanted influenza vaccine which may be administered ≥7 days before or after each study vaccination

  *In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunisation program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its Product Information.
* Concurrently participating in another clinical study, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or medical device)
* Received a vaccine against S. aureus
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions before 2 months after completion of the vaccination series
* History of chronic alcohol consumption and/or drug abuse
* Any study personnel or immediate dependents, family, or household member

All participants at the time of vaccination

* Any clinically significant hematological (hemoglobin level, white blood cell, lymphocyte, neutrophil, eosinophil, platelet count and red blood cell count) and/or biochemical (alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine) laboratory abnormality

Additional exclusion criteria applied only for dose-escalation safety lead-in

* Any active or ongoing illness at screening or time of injection
* History of any serious chronic or progressive disease according to the judgment of the investigator

Additional exclusion criteria applied only for PoP at study entry

* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* Major congenital defects, as assessed by the investigator
* Acute or chronic, clinically significant pulmonary, cardiovascular*, hepatic or renal functional abnormality, neoplasm, diabetes type 1 and uncontrolled diabetes type 2*, as determined by physical examination or laboratory screening tests * Note: Well-controlled type 2 diabetes mellitus (HbA1c <7%) and well-controlled arterial hypertension (blood pressure <140/90 mmHg) can be considered for inclusion in the study.
* Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study
* Individuals at risk for severe or life-threatening SSTIs (e.g., lymphatic or venous insufficiency, liver and kidney disease, IV drug use, etc.)
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study

Additional exclusion criteria applied only for PoP at vaccination

- Microbiological test results of drainage suggest that the SSTI etiology could be other than infection with S. aureus

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKlline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Started (Enrolled set) | 6 | 6 | 6 | 6 | 8 | 105 | 89
Exposed Set (Participants who received at least 1 dose of the study treatment.) | 6 | 6 | 6 | 6 | 8 | 103 | 89
Completed | 6 | 6 | 6 | 6 | 8 | 80 | 79
Not Completed | 0 | 0 | 0 | 0 | 0 | 25 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 20 | 5
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Migrated / Moved from the Study Area | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 105 | 89 | 226
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 6 | 6 | 6 | 6 | 8 | 105 | 89 | 226
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 2 | 6 | 44 | 34 | 99
  Male | 3 | 1 | 1 | 4 | 2 | 61 | 55 | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 5
  Not Hispanic or Latino | 5 | 6 | 6 | 6 | 8 | 66 | 58 | 155
  Not reported | 0 | 0 | 0 | 0 | 0 | 37 | 29 | 66

OUTCOME MEASURES:

1. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With Any and Grade 3 Solicited Administration Site Adverse Events (AEs) After Each Vaccination
Description: The solicited administration site AE(s) assessed are pain, redness and swelling. Any = any solicited administration site AE, regardless of intensity; Grade 3 Pain at injection site = Severe, significant pain at rest, that prevents normal everyday activities; Grade 3 redness/swelling = greater than (>)100 millimeter (mm) diameter.
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-each vaccination; Vaccination 1 on Day 1 and Vaccination 2 on Day 61)
Population: The analysis was performed on Solicited Safety Set (SSS) which included all subjects who received at least 1 dose of the study treatment (Exposed Set) who have solicited safety data. Analysis is presented for Dose-escalation safety lead-in participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Vaccination 1, Pain at injection site, Any | 2 | 3 | 5 | 5 | 1
  Vaccination 1, Pain at injection site, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Redness at injection site, Any | 0 | 1 | 0 | 2 | 0
  Vaccination 1, Redness at injection site, >100 mm | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Swelling at injection site, Any | 0 | 0 | 0 | 1 | 0
  Vaccination 1, Swelling at injection site, >100 mm | 0 | 0 | 0 | 0 | 0
  Vaccination 2, Pain at injection site, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Pain at injection site, Any |  |  |  | 6 | 0
  Vaccination 2, Pain at injection site, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Pain at injection site, Severe |  |  |  | 0 | 0
  Vaccination 2, Redness at injection site, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Redness at injection site, Any |  |  |  | 3 | 0
  Vaccination 2, Redness at injection site, >100 mm: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Redness at injection site, >100 mm |  |  |  | 0 | 0
  Vaccination 2, Swelling at injection site, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Swelling at injection site, Any |  |  |  | 3 | 0
  Vaccination 2, Swelling at injection site, >100 mm: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Swelling at injection site, >100 mm |  |  |  | 0 | 0

2. Primary Outcome: PoP: Number of Participants With Any and Grade 3 Solicited Administration Site AEs After Each Vaccination
Description: The solicited administration site AEs assessed are pain, redness and swelling. Any = any solicited administration site AE, regardless of intensity; Grade 3 Pain at injection site = Severe, significant pain at rest, that prevents normal everyday activities; Grade 3 redness/swelling = greater than (>)100 millimeter (mm) diameter.
Time Frame: as for outcome 1
Population: The analysis was performed on Solicited Safety Set (SSS). Analysis is presented for PoP participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 102 | 88
Participants
  Vaccination 1, Pain at injection site, Any | 56 | 11
  Vaccination 1, Pain at injection site, Severe | 2 | 0
  Vaccination 1, Redness at injection site, Any | 4 | 0
  Vaccination 1, Redness at injection site, >100 mm | 1 | 0
  Vaccination 1, Swelling at injection site, Any | 7 | 1
  Vaccination 1, Swelling at injection site, >100 mm | 2 | 1
  Vaccination 2, Pain at injection site, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Pain at injection site, Any | 42 | 2
  Vaccination 2, Pain at injection site, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Pain at injection site, Severe | 3 | 0
  Vaccination 2, Redness at injection site, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Redness at injection site, Any | 10 | 0
  Vaccination 2, Redness at injection site, >100 mm: number analyzed (Participants) | 66 | 47
  Vaccination 2, Redness at injection site, >100 mm | 4 | 0
  Vaccination 2, Swelling at injection site, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Swelling at injection site, Any | 13 | 0
  Vaccination 2, Swelling at injection site, >100 mm: number analyzed (Participants) | 66 | 47
  Vaccination 2, Swelling at injection site, >100 mm | 3 | 0

3. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With Any and Grade 3 Solicited Systemic AEs After Each Vaccination
Description: The solicited systemic AE(s) assessed are headache, fatigue, nausea, vomiting, diarrhea, abdominal pain, myalgia, shivering and fever. Any = any solicited systemic AE regardless of intensity; Grade 3 headache/fatigue/nausea/abdominal pain/myalgia/shivering = Severe: Prevents daily activity. Grade 3 vomiting = Severe: 6 or more times in 24 hours or requires intravenous hydration. Grade 3 diarrhea = Severe: 6 or more loose stools in 24 hours or requires intravenous hydration. Grade 3 fever = body temperature greater than (>) 40.0°C/104°F.
Time Frame: as for outcome 1
Population: The analysis was performed on Solicited Safety Set (SSS). Analysis is presented for Dose-escalation safety lead-in participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Vaccination 1, Abdominal Pain, Any | 0 | 1 | 0 | 0 | 1
  Vaccination 1, Abdominal Pain, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Diarrhea, Any | 0 | 1 | 1 | 1 | 0
  Vaccination 1, Diarrhea, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Fatigue, Any | 1 | 2 | 3 | 3 | 2
  Vaccination 1, Fatigue, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Fever, Any | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Fever (°C), > 40.0 | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Headache, Any | 0 | 3 | 2 | 1 | 4
  Vaccination 1, Headache, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Myalgia, Any | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Myalgia, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Nausea, Any | 0 | 1 | 2 | 0 | 1
  Vaccination 1, Nausea, Severe | 0 | 0 | 0 | 0 | 1
  Vaccination 1, Shivering, Any | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Shivering, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Vomiting, Any | 0 | 0 | 0 | 0 | 0
  Vaccination 1, Vomiting, Severe | 0 | 0 | 0 | 0 | 0
  Vaccination 2, Abdominal Pain, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Abdominal Pain, Any |  |  |  | 0 | 0
  Vaccination 2, Abdominal Pain, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Abdominal Pain, Severe |  |  |  | 0 | 0
  Vaccination 2, Diarrhea, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Diarrhea, Any |  |  |  | 0 | 0
  Vaccination 2, Diarrhea, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Diarrhea, Severe |  |  |  | 0 | 0
  Vaccination 2, Fatigue, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Fatigue, Any |  |  |  | 5 | 0
  Vaccination 2, Fatigue, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Fatigue, Severe |  |  |  | 1 | 0
  Vaccination 2, Fever, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Fever, Any |  |  |  | 3 | 0
  Vaccination 2, Fever (°C), > 40.0: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Fever (°C), > 40.0 |  |  |  | 0 | 0
  Vaccination 2, Headache, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Headache, Any |  |  |  | 3 | 0
  Vaccination 2, Headache, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Headache, Severe |  |  |  | 1 | 0
  Vaccination 2, Myalgia, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Myalgia, Any |  |  |  | 0 | 0
  Vaccination 2, Myalgia, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Myalgia, Severe |  |  |  | 0 | 0
  Vaccination 2, Nausea, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Nausea, Any |  |  |  | 2 | 0
  Vaccination 2, Nausea, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Nausea, Severe |  |  |  | 0 | 0
  Vaccination 2, Shivering, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Shivering, Any |  |  |  | 0 | 0
  Vaccination 2, Shivering, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Shivering, Severe |  |  |  | 0 | 0
  Vaccination 2, Vomiting, Any: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Vomiting, Any |  |  |  | 0 | 0
  Vaccination 2, Vomiting, Severe: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, Vomiting, Severe |  |  |  | 0 | 0

4. Primary Outcome: PoP: Number of Participants With Any and Grade 3 Solicited Systemic AEs After Each Vaccination
Description: The solicited systemic AE(s) assessed are headache, fatigue, nausea, vomiting, diarrhea, abdominal pain, myalgia, shivering and fever were assessed. Any = any solicited systemic AE regardless of intensity; Grade 3 headache/fatigue/nausea/abdominal pain/myalgia/shivering = Severe: Prevents daily activity. Grade 3 vomiting = Severe: 6 or more times in 24 hours or requires intravenous hydration. Grade 3 diarrhea = Severe: 6 or more loose stools in 24 hours or requires intravenous hydration. Grade 3 fever = body temperature greater than (>) 40.0°C/104°F.
Time Frame: as for outcome 1
Population: The analysis was performed on Solicited Safety Set (SSS). Analysis is presented for PoP participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 102 | 88
Participants
  Vaccination 1, Abdominal Pain, Any | 6 | 6
  Vaccination 1, Abdominal Pain, Severe | 0 | 0
  Vaccination 1, Diarrhea, Any | 11 | 4
  Vaccination 1, Diarrhea, Severe | 0 | 0
  Vaccination 1, Fatigue, Any | 34 | 21
  Vaccination 1, Fatigue, Severe | 2 | 2
  Vaccination 1, Fever, Any | 4 | 1
  Vaccination 1, Fever (°C), > 40.0 | 0 | 0
  Vaccination 1, Headache, Any | 28 | 26
  Vaccination 1, Headache, Severe | 1 | 2
  Vaccination 1, Myalgia, Any | 16 | 10
  Vaccination 1, Myalgia, Severe | 1 | 0
  Vaccination 1, Nausea, Any | 8 | 8
  Vaccination 1, Nausea, Severe | 0 | 0
  Vaccination 1, Shivering, Any | 8 | 5
  Vaccination 1, Shivering, Severe | 0 | 0
  Vaccination 1, Vomiting, Any | 2 | 1
  Vaccination 1, Vomiting, Severe | 0 | 0
  Vaccination 2, Abdominal Pain, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Abdominal Pain, Any | 4 | 0
  Vaccination 2, Abdominal Pain, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Abdominal Pain, Severe | 0 | 0
  Vaccination 2, Diarrhea, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Diarrhea, Any | 4 | 2
  Vaccination 2, Diarrhea, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Diarrhea, Severe | 0 | 0
  Vaccination 2, Fatigue, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Fatigue, Any | 33 | 7
  Vaccination 2, Fatigue, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Fatigue, Severe | 3 | 1
  Vaccination 2, Fever, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Fever, Any | 4 | 1
  Vaccination 2, Fever (°C), > 40.0: number analyzed (Participants) | 66 | 47
  Vaccination 2, Fever (°C), > 40.0 | 0 | 0
  Vaccination 2, Headache, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Headache, Any | 24 | 7
  Vaccination 2, Headache, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Headache, Severe | 3 | 0
  Vaccination 2, Myalgia, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Myalgia, Any | 15 | 2
  Vaccination 2, Myalgia, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Myalgia, Severe | 3 | 0
  Vaccination 2, Nausea, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Nausea, Any | 11 | 4
  Vaccination 2, Nausea, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Nausea, Severe | 1 | 0
  Vaccination 2, Shivering, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Shivering, Any | 11 | 1
  Vaccination 2, Shivering, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Shivering, Severe | 2 | 0
  Vaccination 2, Vomiting, Any: number analyzed (Participants) | 66 | 47
  Vaccination 2, Vomiting, Any | 3 | 0
  Vaccination 2, Vomiting, Severe: number analyzed (Participants) | 66 | 47
  Vaccination 2, Vomiting, Severe | 0 | 0

5. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With Unsolicited AEs (Any, Grade 3, Related, Related Grade 3) After Each Vaccination
Description: An unsolicited adverse event is defined as an adverse event that was not solicited using a Subject Diary and that was spontaneously communicated by a subject who has signed the informed consent. Any unsolicited AE, Grade 3 unsolicited AE, unsolicited AE causally related to the vaccination and Grade 3 unsolicited AE causally related to the vaccination were assessed. A grade 3 AE is an AE that prevents normal, everyday activities.
Time Frame: During 30 days after each vaccination (day of administration and 29 subsequent days post-each vaccination; Vaccination 1 on Day 1 and Vaccination 2 on Day 61)
Population: The analysis was performed on the Unsolicited Safety Set (USS) which included all subjects who received at least 1 dose of the study treatment (Exposed Set) that report unsolicited AEs/report not having unsolicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  Vaccination 1, At least one unsolicited adverse event | 1 | 3 | 1 | 0 | 0
  Vaccination 1, At least one related unsolicited adverse event | 1 | 2 | 0 | 0 | 0
  Vaccination 1, At least one grade 3 unsolicited adverse event | 0 | 0 | 0 | 0 | 0
  Vaccination 1, At least one grade 3 related unsolicited adverse event | 0 | 0 | 0 | 0 | 0
  Vaccination 2, At least one unsolicited adverse event: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, At least one unsolicited adverse event |  |  |  | 2 | 0
  Vaccination 2, At least one related unsolicited adverse event: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, At least one related unsolicited adverse event |  |  |  | 2 | 0
  Vaccination 2, At least one grade 3 unsolicited adverse event: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, At least one grade 3 unsolicited adverse event |  |  |  | 0 | 0
  Vaccination 2, At least one grade 3 related unsolicited adverse event: number analyzed (Participants) | 0 | 0 | 0 | 6 | 2
  Vaccination 2, At least one grade 3 related unsolicited adverse event |  |  |  | 0 | 0

6. Primary Outcome: PoP: Number of Participants With Unsolicited AEs (Any, Grade 3, Related, Related Grade 3) After Each Vaccination
Description: as for outcome 5
Time Frame: as for outcome 5
Population: The analysis was performed on USS.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 103 | 89
Participants
  Vaccination 1, At least one unsolicited adverse event | 32 | 26
  Vaccination 1, At least one related unsolicited adverse event | 16 | 4
  Vaccination 1, At least one grade 3 unsolicited adverse event | 0 | 1
  Vaccination 1, At least one grade 3 related unsolicited adverse event | 0 | 0
  Vaccination 2, At least one unsolicited adverse event: number analyzed (Participants) | 67 | 48
  Vaccination 2, At least one unsolicited adverse event | 23 | 7
  Vaccination 2, At least one related unsolicited adverse event: number analyzed (Participants) | 67 | 48
  Vaccination 2, At least one related unsolicited adverse event | 12 | 4
  Vaccination 2, At least one grade 3 unsolicited adverse event: number analyzed (Participants) | 67 | 48
  Vaccination 2, At least one grade 3 unsolicited adverse event | 1 | 1
  Vaccination 2, At least one grade 3 related unsolicited adverse event: number analyzed (Participants) | 67 | 48
  Vaccination 2, At least one grade 3 related unsolicited adverse event | 1 | 1

7. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With Serious AEs (SAEs) up to 1 Year Post First Vaccination
Description: A SAE is defined as any untoward medical occurrence that, at any dose: resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment. A grade 3 SAE is a SAE that prevents normal, everyday activities.
Time Frame: From Day 1 to Day 366
Population: The analysis was performed on the Exposed Set (ES) that included all subjects who received at least 1 dose of the study treatment. The allocation in a group is done in function of the administered treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants
  At least one SAE | 0 | 0 | 0 | 0 | 0
  At least one serious related AE | 0 | 0 | 0 | 0 | 0
  Any Grade 3 SAE | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With SAEs up to 1 Year Post Second Vaccination
Description: as for outcome 7
Time Frame: From Day 61 to Day 426 (post vaccination at Day 61)
Population: The analysis was performed on ES. Only participants that received a second vaccination on Day 61 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 2
Participants
  At least one SAE | 0 | 0
  At least one serious related AE | 0 | 0
  Any Grade 3 SAE | 0 | 0

9. Primary Outcome: PoP: Number of Participants With SAEs
Description: as for outcome 7
Time Frame: From Day 1 to Day 426
Population: The analysis was performed on ES. The allocation in a group is done in function of the administered treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 103 | 89
Participants
  At least one SAE | 5 | 5
  At least one serious related AE | 0 | 0
  Any Grade 3 SAE | 3 | 2

10. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With Potential Immune-mediated Diseases (pIMDs) up to 1 Year Post First Vaccination
Description: pIMDs are defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 1 to Day 366
Population: The analysis was performed on ES.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Dose-escalation Safety lead-in: Number of Participants With pIMDs up to 1 Year Post Second Vaccination
Description: as for outcome 10
Time Frame: From Day 61 to Day 426 (post vaccination at Day 61)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo
Number analyzed (Participants) | 6 | 2
Participants | 0 | 0

12. Primary Outcome: PoP: Number of Participants With Potential Immune-mediated Diseases (pIMDs)
Description: as for outcome 10
Time Frame: From Day 1 to Day 426
Population: The analysis was performed on ES.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 103 | 89
Participants | 0 | 0

13. Primary Outcome: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Haematological and Biochemical Laboratory Parameters
Description: The Biochemical parameters assessed were: Creatinine, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and the Haematological parameters assessed were: Haemoglobin, white blood cells (WBC) decrease, WBC increase, Neutrophils decrease, Platelets decrease, Lymphocytes decrease, Eosinophils increase. Hematological and biochemical laboratory results are defined as follows: <parameter>,<grade at baseline>,<grade at visit> (e.g. ALT, Grade 0, Grade 0), where Grade 0 = a non-missing parameter value for which grade could not be derived according to the grading scale and does not belong to Grade 1-4; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life-Threatening. Grading following the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007). Unknown = parameter value missing for the specified parameter.
Time Frame: On Day 8 compared to Baseline (Day 1)
Population: The analysis was performed on the Laboratory Safety Set that was a subset of the Unsolicited Safety Set. Only participants that had available data as per pre-assigned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 8 | 29 | 11
Participants
  ALT, Grade 0, Grade 0 | 6 | 6 | 4 | 5 | 8 | 26 | 11
  ALT, Grade 1, Grade 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  ALT, Grade 1, Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  AST, Grade 0, Grade 0 | 6 | 6 | 5 | 5 | 8 | 28 | 11
  AST, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AST, Grade 1, Grade 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine, Unknown, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine, Grade 0, Grade 0 | 6 | 6 | 5 | 6 | 8 | 29 | 10
  Eosinophils Increase, Grade 0, Grade 0 | 6 | 6 | 5 | 6 | 8 | 27 | 10
  Eosinophils Increase, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Eosinophils Increase, Grade 1, Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Haemoglobin Decrease, Grade 0, Grade 0 | 6 | 5 | 4 | 6 | 8 | 20 | 10
  Haemoglobin Decrease, Grade 0, Grade 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1
  Haemoglobin Decrease, Grade 1, Grade 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Haemoglobin Decrease, Grade 1, Grade 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0
  Lymphocytes Decrease, Grade 0, Grade 0 | 6 | 6 | 4 | 6 | 8 | 29 | 11
  Lymphocytes Decrease, Grade 1, Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils Decrease, Grade 0, Grade 0 | 6 | 6 | 5 | 6 | 7 | 29 | 11
  Neutrophils Decrease, Grade 0, Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets Decrease, Grade 0, Grade 0 | 6 | 6 | 5 | 6 | 8 | 29 | 11
  WBC Decrease, Grade 0, Grade 0 | 6 | 6 | 5 | 6 | 8 | 29 | 11
  WBC Increase, Grade 0, Grade 0 | 6 | 5 | 4 | 6 | 7 | 26 | 11
  WBC Increase, Grade 0, Grade 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  WBC Increase, Grade 1, Grade 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0

14. Primary Outcome: Number of Participants With Maximum Toxicity Grade Increase From Baseline for Haematological and Biochemical Laboratory Parameters
Description: The Biochemical parameters assessed were: Creatinine, AST, ALT and the Haematological parameters assessed were: Haemoglobin, WBC decrease, WBC increase, Neutrophils decrease, Platelets decrease, Lymphocytes decrease, Eosinophils increase. Hematological and biochemical laboratory results are defined as follows: <parameter>,<grade at baseline>,<grade at visit> (e.g. ALT, Grade 0, Grade 0), where Grade 0 = a non-missing parameter value for which grade could not be derived according to the grading scale and does not belong to Grade 1-4; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life-Threatening. Grading following the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007). Unknown = parameter value missing for the specified parameter.
Time Frame: On Day 68 compared to Baseline (Day 61)
Population: The analysis was performed on the Laboratory Safety Set. Only participants that had available data as per pre-assigned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 6 | 2 | 28 | 11
Participants
  ALT, Unknown, Grade 0 | 0 | 0 | 1 | 0
  ALT, Grade 0, Grade 0 | 6 | 2 | 26 | 11
  ALT, Grade 1, Grade 1 | 0 | 0 | 1 | 0
  AST, Unknown, Grade 0 | 0 | 0 | 1 | 0
  AST, Grade 0, Grade 0 | 6 | 2 | 26 | 10
  AST, Grade 0, Grade 1 | 0 | 0 | 1 | 0
  AST, Grade 1, Grade 0 | 0 | 0 | 0 | 1
  Creatinine, Unknown, Grade 0 | 0 | 0 | 1 | 0
  Creatinine, Grade 0, Grade 0 | 6 | 2 | 27 | 11
  Eosinophils Increase, Unknown, Grade 0 | 1 | 0 | 1 | 0
  Eosinophils Increase, Grade 0, Grade 0 | 5 | 2 | 25 | 10
  Eosinophils Increase, Grade 0, Grade 1 | 0 | 0 | 1 | 0
  Eosinophils Increase, Grade 1, Grade 1 | 0 | 0 | 1 | 1
  Haemoglobin Decrease, Unknown, Grade 0 | 1 | 0 | 1 | 0
  Haemoglobin Decrease, Grade 0, Grade 0 | 5 | 2 | 21 | 9
  Haemoglobin Decrease, Grade 0, Grade 1 | 0 | 0 | 2 | 0
  Haemoglobin Decrease, Grade 1, Grade 0 | 0 | 0 | 2 | 0
  Haemoglobin Decrease, Grade 1, Grade 1 | 0 | 0 | 1 | 2
  Haemoglobin Decrease, Grade 1, Grade 2 | 0 | 0 | 1 | 0
  Lymphocytes Decrease, Unknown, Grade 0 | 1 | 0 | 1 | 0
  Lymphocytes Decrease, Grade 0, Grade 0 | 5 | 2 | 26 | 11
  Lymphocytes Decrease, Grade 0, Grade 1 | 0 | 0 | 1 | 0
  Neutrophils Decrease, Unknown, Grade 0 | 1 | 0 | 1 | 0
  Neutrophils Decrease, Grade 0, Grade 0 | 5 | 2 | 25 | 11
  Neutrophils Decrease, Grade 1, Grade 0 | 0 | 0 | 1 | 0
  Neutrophils Decrease, Grade 1, Grade 1 | 0 | 0 | 1 | 0
  Platelets Decrease, Unknown, Grade 0 | 1 | 0 | 1 | 0
  Platelets Decrease, Grade 0, Grade 0 | 5 | 2 | 27 | 11
  WBC Decrease, Unknown, Grade 0 | 1 | 0 | 1 | 0
  WBC Decrease, Grade 0, Grade 0 | 5 | 2 | 26 | 11
  WBC Decrease, Grade 1, Grade 0 | 0 | 0 | 1 | 0
  WBC Increase, Unknown, Grade 0 | 1 | 0 | 1 | 0
  WBC Increase, Grade 0, Grade 0 | 5 | 2 | 25 | 10
  WBC Increase, Grade 0, Grade 1 | 0 | 0 | 1 | 1
  WBC Increase, Grade 1, Grade 0 | 0 | 0 | 1 | 0

15. Primary Outcome: Number of Participants With Haematological and Biochemical Laboratory Change From Baseline Values
Description: The Biochemical parameters assessed were: Creatinine, AST, ALT and the Haematological parameters assessed were: Haemoglobin, WBC decrease, WBC increase, Neutrophils decrease, Platelets decrease, Lymphocytes decrease, Eosinophils increase. Hematological and biochemical laboratory results are defined as follows: <parameter>,<any grade at baseline>,<grade at visit> (e.g. ALT, Any, Grade 0), where Grade 0 = a non-missing parameter value for which grade could not be derived according to the grading scale and does not belong to Grade 1-4; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life-Threatening. Grading following the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007). Unknown = parameter value missing for the specified parameter.
Time Frame: On Day 8
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 8 | 29 | 11
Participants
  ALT, Any, Grade 0 | 6 | 6 | 5 | 6 | 8 | 27 | 11
  ALT, Any, Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  AST, Any, Grade 0 | 6 | 6 | 5 | 6 | 8 | 28 | 11
  AST, Any, Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine, Any, Grade 0 | 6 | 6 | 5 | 6 | 8 | 29 | 11
  Eosinophils Increase, Any, Grade 0 | 6 | 6 | 5 | 6 | 8 | 27 | 11
  Eosinophils Increase, Any, Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Haemoglobin Decrease, Any, Grade 0 | 6 | 5 | 4 | 6 | 8 | 22 | 10
  Haemoglobin Decrease, Any, Grade 1 | 0 | 1 | 1 | 0 | 0 | 7 | 1
  Lymphocytes Decrease, Any, Grade 0 | 6 | 6 | 4 | 6 | 8 | 29 | 11
  Lymphocytes Decrease, Any, Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils Decrease, Any, Grade 0 | 6 | 6 | 5 | 6 | 7 | 29 | 11
  Neutrophils Decrease, Any, Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets Decrease, Any, Grade 0 | 6 | 6 | 5 | 6 | 8 | 29 | 11
  WBC Decrease, Any, Grade 0 | 6 | 6 | 5 | 6 | 8 | 29 | 11
  WBC Increase, Any, Grade 0 | 6 | 5 | 5 | 6 | 8 | 27 | 11
  WBC Increase, Any, Grade 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0

16. Primary Outcome: Number of Participants With Haematological and Biochemical Laboratory Change From Baseline Values
Description: as for outcome 15
Time Frame: On Day 68
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 6 | 2 | 28 | 11
Participants
  ALT, Any, Grade 0 | 6 | 2 | 27 | 11
  ALT, Any, Grade 1 | 0 | 0 | 1 | 0
  AST, Any, Grade 0 | 6 | 2 | 27 | 11
  AST, Any, Grade 1 | 0 | 0 | 1 | 0
  Creatinine, Any, Grade 0 | 6 | 2 | 28 | 11
  Eosinophils Increase, Any, Grade 0 | 6 | 2 | 26 | 10
  Eosinophils Increase, Any, Grade 1 | 0 | 0 | 2 | 1
  Haemoglobin Decrease, Any, Grade 0 | 6 | 2 | 24 | 9
  Haemoglobin Decrease, Any, Grade 1 | 0 | 0 | 3 | 2
  Haemoglobin Decrease, Any, Grade 2 | 0 | 0 | 1 | 0
  Lymphocytes Decrease, Any, Grade 0 | 6 | 2 | 27 | 11
  Lymphocytes Decrease, Any, Grade 1 | 0 | 0 | 1 | 0
  Neutrophils Decrease, Any, Grade 0 | 6 | 2 | 27 | 11
  Neutrophils Decrease, Any, Grade 1 | 0 | 0 | 1 | 0
  Platelets Decrease, Any, Grade 0 | 6 | 2 | 28 | 11
  WBC Decrease, Any, Grade 0 | 6 | 2 | 28 | 11
  WBC Increase, Any, Grade 0 | 6 | 2 | 27 | 10
  WBC Increase, Any, Grade 1 | 0 | 0 | 1 | 1

17. Secondary Outcome: Number of Participants With at Least One Culture Confirmed Case of Recurrent Staphylococcus Aureus (S. Aureus) Skin and Soft Tissue Infection (SSTI) - Interim Analysis
Description: An interim analysis was performed after 13 cases of recurrent SA-SSTI were reported following 14 days from the study intervention dose 2.
Time Frame: From Day 75 to Day 426
Population: The analysis was performed on Interim analysis Proof of Principle (PoP) - modified Full Analysis Set (mFAS) which included all subjects who received full study treatment course to which they are randomised and have post-vaccination efficacy data.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 38 | 21
Participants | 10 | 3
Statistical Analysis 1: Comparison: Proof of Principle (PoP): Full Dose Adj vs PoP: Placebo; Test type: Superiority; p = 0.8042, Log Rank; One-sided Group Sequential Design with non-binding beta, yielding two CIs based on cumulative alpha (92.5%) and beta (80.5%) spending; Vaccine Efficacy (VE) = -74.76, 92.5% CI [-680.61 to 36.62] — Vaccine Efficacy (VE) is defined as 1 minus the hazard ratio times 100

18. Secondary Outcome: Number of Participants With at Least One Culture Confirmed Case of Recurrent S. Aureus SSTI - Final Analysis
Description: After encountering futility at the interim analysis, an EOS analysis was conducted when at least one culture-confirmed case of recurrent SA-SSTI was identified 14 days after the second dose of the vaccine. For the final analysis, all the data collected by End of Study (EoS; Last Participant Last Visit) were analyzed for descriptive purposes.
Time Frame: From Day 75 to Day 426
Population: The analysis was performed on EoS analysis PoP mFAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 66 | 48
Participants | 14 | 8
Statistical Analysis 1: Comparison: Proof of Principle (PoP): Full Dose Adj vs PoP: Placebo; Test type: Other; Vaccine Efficacy (VE) = -38.09, 95% CI 2-sided [-245.77 to 40.86] — Vaccine Efficacy (VE) is defined as 1 minus the hazard ratio times 100

19. Secondary Outcome: Number of Participants With at Least One Culture Confirmed Case of Recurrent S. Aureus SSTI - Final Analysis
Description: An EOS analysis was conducted when at least one culture-confirmed case of recurrent SA-SSTI was identified 14 days after the first dose of the vaccine. For the final analysis, all the data collected by End of Study (EoS; Last Participant Last Visit) were analyzed for descriptive purposes.
Time Frame: From Day 15 to Day 426
Population: The analysis was performed on the EOS PoP: Full Analysis Set (FAS) which included all subjects who received at least 1 dose of the study treatment and have post-vaccination efficacy data.
Measure: Count of Participants; unit: Participants
Arm/Group | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
Number analyzed (Participants) | 103 | 89
Participants | 18 | 10
Statistical Analysis 1: Comparison: Proof of Principle (PoP): Full Dose Adj vs PoP: Placebo; Test type: Other; Vaccine Efficacy (VE) = -75.52, 95% CI 2-sided [-295.41 to 17.46] — Vaccine Efficacy (VE) is defined as 1 minus the hazard ratio times 100

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7 (post vaccination 1) and from Day 61 to Day 67 (post Vaccination 2 only for Group 4 and PoP epoch). Unsolicited AEs were collected from Day 1 to Day 30 (post vaccination 1) and from Day 61 to Day 90 (post vaccination 2 only for Group 4 and PoP epoch). SAEs and pIMDs were collected from Day 1 to Day 366 (post vaccination 1, dose escalation), Day 61 to Day 426 (post vaccination 2, only for Group 4), from Day 1 to Day 426 for PoP epoch
Description: Adverse events are reported on the Exposed Set, who received at least 1 dose of the study treatment.
Arm/Group | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj | Dose-escalation Safety Lead-in Epoch: Placebo | Proof of Principle (PoP): Full Dose Adj | PoP: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/103 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 5/103 | 5/89
Other Adverse Events (participants affected / at risk) | 3/6 | 6/6 | 5/6 | 6/6 | 5/8 | 82/103 | 60/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) (N=6) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj (N=6) | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj (N=6) | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj (N=6) | Dose-escalation Safety Lead-in Epoch: Placebo (N=8) | Proof of Principle (PoP): Full Dose Adj (N=103) | PoP: Placebo (N=89)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Dose-escalation Safety Lead-in Epoch: Half Dose Non-Adjuvant (Non-Adj) (N=6) | Group 2 Dose-escalation Safety Lead-in Epoch: Full Dose Non-Adj (N=6) | Group 3 Dose-escalation Safety Lead-in Epoch: Half Dose Adj (N=6) | Group 4 Dose-escalation Safety Lead-in Epoch: Full Dose Adj (N=6) | Dose-escalation Safety Lead-in Epoch: Placebo (N=8) | Proof of Principle (PoP): Full Dose Adj (N=103) | PoP: Placebo (N=89)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (12) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 14 (17) | 4 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 18 (23) | 10 (12)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 20 (22) | 6 (6)
Fatigue (General disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (8) | 2 (2) | 46 (70) | 24 (29)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 12 (16) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site macule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 4 (4) | 5 (5) | 6 (13) | 1 (1) | 65 (114) | 13 (14)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 16 (23) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 12 (12) | 3 (3)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin graft failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 27 (32) | 10 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (4) | 4 (4) | 40 (58) | 28 (37)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04420221/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT04420221/SAP_001.pdf